CLINICAL TRIAL: NCT04787367
Title: Laparoscopic TAP Block for Sleeve Gastrectomy: Does Timing Matter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarah Diaz (Other)
Responsible Party: Sponsor-Investigator, Sarah Diaz, Sub-Investigator, Henry Ford Health System
Organization: Henry Ford Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 643256
Record Dates: First submitted 2018-05-08; First posted 2021-03-08 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Pain, Postoperative
Keywords: TAP block; Obesity; Sleeve gastrectomy; Bariatrics; Post-operative pain
MeSH Terms: conditions — Obesity; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is a single blinded, prospective study designed to determine optimal timing of TAP block in laparoscopic gastric sleeve patients. Patients will randomly be assigned to the early intra-operative TAP block group or the late intra-operative TAP block group.
Who Masked: Participant
Masking Description: The patient will be unaware of when they received the block. The nursing assistants checking the pain score will also be unaware of the timing of the block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early-operative TAP block (Experimental): The TAP block will be administered after the placement of the camera port.
  Interventions: Procedure: TAP block
- Late-operative TAP block (Experimental): The TAP block will be administered at the completion of the case just before removing the camera port.
  Interventions: Procedure: TAP block

INTERVENTIONS:
Procedure: TAP block — An 18-gauge needle will be introduced externally at the center of the mid axillary line between the lower costal margin and the iliac crest until the surgeon feels a "pop," after which the surgeon will inject the first 2 mL of 0.25% bupivicaine to verify the correct position. Doyle's internal bulge sign (the bulge seen when the transversus abdominis muscle and peritoneum is pushed internally) will be visualized and the remainder of the 60 mL of 0.25% bupivacaine will be injected. The contralateral block will be performed according to the same technique but with only 30 ml of bupivicaine.

SUMMARY:
The goal of this study is to investigate whether an early intraoperative transverse abdominis plane block (TAP block) will provide superior analgesia to a late intraoperative TAP block. A fixed amount of bupivacaine will be used for the TAP block and the primary outcomes will be measured by patient reported numerical assessment scores for pain.

DETAILED DESCRIPTION:
This is a single blinded, prospective study designed to determine optimal timing of transverse abdominis plane block (TAP block) in laparoscopic gastric sleeve patients. Research has shown that administration of TAP block during these cases does show improved post-operative pain control. There are no trials specifically evaluating the timing of administration in regards to superiority of pain control. To the investigators knowledge, no prospective study has ever been done investigating whether TAP block performed at the beginning of the case versus at the end of the case makes a difference in the amount of relief experienced by the patient. the investigators hypothesize that early intra-operative block will be superior to late intra-operative block in both post-operative pain as well as decreased length of stay in hospital secondary to reduction in peripheral and central nervous system hyper excitability. Before beginning the research study, ~200 plain envelopes will be made each containing one option written on paper indicating early intra-operative or late intra-operative TAP block. There will be equal numbers of both options. It will be the responsibility of either the PI or sub-investigators to select a random envelope and bring it to the operating room at the time of surgery. All patients involved in the study will have given informed consent in the office prior to surgery. On the day of surgery after the patient is induced and intubated, the PI or sub-investigator will open the envelope revealing the timing of the TAP block. Depending on what is revealed from the envelope, the patient will either receive the early intra-operative TAP block or the late intra-operative TAP block. The TAP block will be performed using 60 ml for right sided TAP block (side of specimen extraction) and 30 ml for left sided TAP block (non extraction side). 30 ml of bupivicaine solution will also be used for intraperitoneal irrigation as is already routinely done during these cases by the primary surgeon for additional analgesia. This will be performed at the conclusion of all cases regardless of which arm the patient is in. For the early intra-operative TAP block, optiview trocar entrance will be performed in the upper abdomen followed by CO2 insufflation. After introduction of the camera into this trocar, the right lateral abdominal wall will be visualized with the laparoscope. An 18-gauge needle will be introduced externally at the center of the mid axillary line between the lower costal margin and the iliac crest until the surgeon feels a "pop," after which the surgeon will inject the first 2 mL of 0.25% bupivicaine to verify the correct position. Doyle's internal bulge sign (the bulge seen when the transversus abdominis muscle and peritoneum is pushed internally) will be visualized and the remainder of the 60 mL of 0.25% bupivacaine will be injected. The contralateral block will be performed according to the same technique but with only 30 ml of bupivicaine. The late post-operative block will be performed in the same fashion but after completion of the surgery just prior to removing the trocars and desufflation. The intraperitoneal irrigation with 0.25% bupivicaine solution will be performed at the end of the case using 30 ml total sprayed above the stomach, under the diaphragm, and over the bed of the spleen. All other medications intra-op and post-op including anesthesia will remain standardized according to the current HF Macomb bariatrics protocols. The data collection will take place immediately post-op, 4, 8, 12, 16, 20, and 24 hours post-op using the numerical assessment score (NAS) for pain which will be performed at the time vitals are taken by the nursing aids. The investigators will also be analyzing post-operative vomiting and length of stay in hours.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing laparoscopic sleeve gastrectomy

Exclusion Criteria:

* Conversion to open procedure
* Prior history of narcotic use (which will be defined as any narcotics used on a recreational basis or any narcotic used for pain relief without having had recent operation or injury)
* Current narcotic use at time of surgery
* Prolonged case time defined as >1 standard deviation over average time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Patient reported pain | Immediately post-operatively (upon arrival to PACU). These pain scales will be done by nurses/nursing aids taking vitals.
  Using the numerical assessment system, the patient will report their pain by choosing a number 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, or 10. On the scale, 0 means no pain (best outcome) and 10 means the most pain (worst outcome). The patients will identify where on the spectrum their pain lays prior to receiving any possible pain medication.The pain scores will be averaged within the two groups at each time interval collected.
Patient reported pain | 4 hours post-operatively. These pain scales will be done by nurses/nursing aids taking vitals.
  Using the numerical assessment system, the patient will report their pain by choosing a number 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, or 10. On the scale, 0 means no pain (best outcome) and 10 means the most pain (worst outcome). The patients will identify where on the spectrum their pain lays prior to receiving any possible pain medication.The pain scores will be averaged within the two groups at each time interval collected.
Patient reported pain | 8 hours post-operatively. These pain scales will be done by nurses/nursing aids taking vitals.
  Using the numerical assessment system, the patient will report their pain by choosing a number 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, or 10. On the scale, 0 means no pain (best outcome) and 10 means the most pain (worst outcome). The patients will identify where on the spectrum their pain lays prior to receiving any possible pain medication.The pain scores will be averaged within the two groups at each time interval collected.
Patient reported pain | 12 hours post-operatively. These pain scales will be done by nurses/nursing aids taking vitals.
  Using the numerical assessment system, the patient will report their pain by choosing a number 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, or 10. On the scale, 0 means no pain (best outcome) and 10 means the most pain (worst outcome). The patients will identify where on the spectrum their pain lays prior to receiving any possible pain medication.The pain scores will be averaged within the two groups at each time interval collected.
Patient reported pain | 16 hours post-operatively. These pain scales will be done by nurses/nursing aids taking vitals.
  Using the numerical assessment system, the patient will report their pain by choosing a number 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, or 10. On the scale, 0 means no pain (best outcome) and 10 means the most pain (worst outcome). The patients will identify where on the spectrum their pain lays prior to receiving any possible pain medication.The pain scores will be averaged within the two groups at each time interval collected.
Patient reported pain | 20 hours post-operatively. These pain scales will be done by nurses/nursing aids taking vitals.
  Using the numerical assessment system, the patient will report their pain by choosing a number 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, or 10. On the scale, 0 means no pain (best outcome) and 10 means the most pain (worst outcome). The patients will identify where on the spectrum their pain lays prior to receiving any possible pain medication.The pain scores will be averaged within the two groups at each time interval collected.
Patient reported pain | 24 hours post-operatively. These pain scales will be done by nurses/nursing aids taking vitals.
  Using the numerical assessment system, the patient will report their pain by choosing a number 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, or 10. On the scale, 0 means no pain (best outcome) and 10 means the most pain (worst outcome). The patients will identify where on the spectrum their pain lays prior to receiving any possible pain medication.The pain scores will be averaged within the two groups at each time interval collected.

SECONDARY OUTCOMES:
Length of stay | Day of surgery to day of discharge up to 30 days
  Days spent in hospital including day of surgery
Narcotic use | Starting with administration of opioid medication in PACU until time of discharge up to 30 days
  We will measure the amount of opioid medication given to the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Carlin, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Macomb Hospital, Clinton Township, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT04787367/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT04787367/ICF_001.pdf